CLINICAL TRIAL: NCT06605014
Title: Characterization of Somatic Dysfunction in Patients With Acute Cerebrovascular Disease
Brief Title: Somatic Dysfunction in Patients With Acute Cerebrovascular Disease
Acronym: SOMADC-AC
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Other Study IDs: 1901775; 23151879 (Other Grant/Funding Number: American Osteopathic Association)
Record Dates: First submitted 2024-07-25; First posted 2024-09-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Stroke, Acute; TIA; Reproducibility of Results; Osteopathic Manipulation; Health-Related Quality-of-Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SOMADC-AC Cohort: 1. Asymptomatic adult volunteers
  2. Patients admitted with TIA
  3. Patients admitted with acute ischemic stroke

SUMMARY:
The goals of this observational study are to test the reliability of a new, standardized physical examination method to identify motion problems within joints or groups of joints among adult asymptomatic volunteers and in patients hospitalized with stroke or stroke-like episodes (e.g., transient ischemic attack, TIA). The main questions this investigation aims to answer are:

* Can different, independent providers reliability quantify motion pattern problems using a systematic approach called, The Functional Pathology of the Musculoskeletal System (FPMSS) model?
* Are there differences in joint(s) motion patterns among asymptomatic volunteers, patients with TIA (people with brain disease without new neurologic disability), and recent ischemic stroke (patients with new stroke-related-disability, e.g., paralysis)?
* Is there an association between joint(s) motion impairment severity and stroke survivor outcomes?

Participants (asymptomatic and those with stroke) will undergo a set of repeated paired, musculoskeletal physical exams by independent providers blinded to each other's assessments and patient information. Researchers will compare the severity, location, and quantity of joint(s) motion impairment between these three groups with the physical examination methodology (FPMSS). Clinical information (e.g., test results, diagnoses, brain imaging, medical history) will be collected from patients admitted for TIA and stroke. Enrolled participants with recent stroke will complete a survey three months after hospitalization to determine their self-perceived quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18 years

Admission diagnosis:

* ischemic stroke OR
* transient ischemic attack (TIA). A prior history of TIA but without stroke may be enrolled.
* Neurologic stability or lack of significant deterioration (i.e. ∆ NIHSS<4) for at least 24 hours (defined by clinical documentation and/or communication with provider team(s)) in stroke subjects
* Able to sit upright, lie supine, and when able lateral recumbent left/right positions with assist independently or with minimal person assist
* Anticipated length of stay greater > or = 2 days for ischemic stroke. TIA patients average length of stay is < 2 days, and can be enrolled in the study.

Exclusion Criteria:

* Acute skeletal fracture or known dislocation; history of pathologic (osteoporotic or neoplastic) skeletal fracture of thoracic cage, hip/pelvis/sacrum, or vertebral column
* Prior history of ICH, ischemic stroke, confirmed by imaging and/or clinical evaluation. Patients with imaging showing "chronic stroke" who have never received a diagnosis of stroke and/or have not been previously symptomatic may still be enrolled, based on the Investigator's clinical judgement.
* Spinal column support brace (e.g. cervical collar)
* Anticipated neurosurgical intervention during hospitalization: decompressive hemicraniectomy, hematoma evacuation (defined by clinical documentation and/or communication with provider team(s))
* Current endotracheal intubation (*note: extubated patients can be evaluated for eligibility)
* History of spinal cord injury with residual neuromuscular or sensory disability
* History of recent trauma within the past 30 days
* Known ligament, musculotendinous, or bone lesion
* Clinical condition that would interfere with execution of movement or palpatory diagnostic testing, e.g. chronic pain
* History of spinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 Asymptomatic adult volunteers (e.g., medical center employees) will be recruited to undergo paired, repeated osteopathic physical examinations and serve as controls.
  20 disease controls (TIA) will undergo a single paired assessment by two independent raters
  80 patients recently admitted with acute ischemic stroke will undergo repeated paired independent rater assessments throughout hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Examiner Rater-Reliability | 3 to 14 days
  Test intra- and inter-rater reliability in identifying osteopathic somatic dysfunction (joint(s) motion impairment) among asymptomatic volunteers, patients with TIA, and recently admitted patients with stroke.
Functional Pathology of the Musculoskeletal System | 3-14 days
  A total of 80 specific musculoskeletal examination tests are performed assessing the amount of available motion in the spine, upper extremities, lower extremities, and pelvis. Navigational Motions (i.e., whole upper limb motion at shoulder) are scored on a scale of 1-4 with one representing the least loss of motion and 4 representing the most and Component Motions (i.e., motion of foot at ankle) scored on a scale of 0-3 with 0 representing "normal motion" and 3 representing "no motion".
National Institutes of Health Neuro-Quality of Life (QoL) survey | 90 days
  Quantify self-reported health-related quality-of-life (QoL) 90 days after ischemic stroke. Patient response domain scores have a normative distribution and are compared against general population means (50, with a standard deviation of 10; range 10-90). Interpreting value responses above or below means are based on the specific questions - i.e., higher scores do not uniformly reflect improvement while lower scores do not necessarily reflect poorer status. Patient will receive a digitally distributed survey inquiring about QoL domains surrounding mobility, satisfaction with and ability to participate in social roles, mood, fatigue, anxiety, cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Yee, D.O., Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States